CLINICAL TRIAL: NCT02304718
Title: Cycle Study:an Exercise Intervention to Prevent Gestational Diabetes in Overweight and Obese Chinese Pregnant Women
Brief Title: Exercise Intervention to Prevent Gestational Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Wang Chen, Ms, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 400010558
Record Dates: First submitted 2014-11-24; First posted 2014-12-02 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-08

CONDITIONS: Gestational Diabetes Mellitus
Keywords: GDM; pregnancy outcome; obesity; exercise; overweight
MeSH Terms: conditions — Diabetes, Gestational; Obesity; Motor Activity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- exercise intervention group (Experimental): Pregnant women randomised to the exercise intervention group will complete three supervised, exercise sessions each week, exercise sessions completed on alternate days, and lasts until they give birth by using a stational bike. And also they will have regular prenatal care.
  Interventions: Behavioral: Stationary bike
- control group (No Intervention): Pregnant women randomised to the control group only have regular prenatal care.

INTERVENTIONS:
Behavioral: Stationary bike
  Arms: exercise intervention group

SUMMARY:
This study evaluates the role of exercise intervention in reducing the risk of gestational diabetes mellitus(GDM) risk of overweight/obese(prepregnancy BMI≥24kg/m^2） Chinese pregnant women. Half of participants will have exercise intervention, while the other half will not. Both of the two group will have regular prenatal care.

DETAILED DESCRIPTION:
An increasing number of women are entering pregnancy in an overweight or obese state. The overweight/obesity epidemic among women of reproductive age has led to an increasing incidence of gestational diabetes mellitus (GDM)，and other metabolic and obstetric complications, such as fetal macrosomia, maternal obesity and type 2 diabetes.

Exercise may be a non-invasive therapeutic option for preventing and managing GDM that can be readily applied to the antenatal population.But so far, the effects of exercise interventions on the incidence of GDM and other adverse perinatal outcomes have been scarce, especially in Chinese pregnant women.

So the aim of the investigators study is to evaluate whether exercise intervention in overweight/obese(prepregnancy BMI≥24kg/m^2） Chinese pregnant women can reduce their risk of GDM and GDM related adverse pregnant outcomes.

Overweight/obese Chinese pregnant women (prepregnancy BMI≥24kg/m^2） will be randomly divided into exercise intervention group and control group in their first trimester（less than 13 gestational weeks), pregnant women randomised to the exercise intervention group will complete three supervised, exercise sessions each week by using a stational bike, and exercise sessions will be completed on alternate days. Both exercise group and control group have regular prenatal care.

During 24-28 gestatioanl weeks,GDM will be diagnosed by an oral glucose tolerance test (OGTT) according to the new World Health Organization criteria as fasting glucose level in fasting whole blood 5.1 mmol/L or more, or 2-hour value 8.5mmol/L or more.Then the investigators can compare the GDM risk in each group, and find out if exercise intervention can reduce the risk of GDM in overweight/obese Chinese pregnant women.

Following，no matter pregnant women who were diagnosed with GDM in the intervention group or the control group,they will all have standard medical managemen, and continue what they do before until they give birth. That means pregnnat women in the intervention group will continue to have exercise intervention and regular prenatal care despite whether they have GDM or not.

So when they give birth, the investigators can compare pregnant outcomes between four groups, that is exercise group without GDM, exercise group with GDM, control group without GDM and control group with GDM.And the pregnant outcomes include preterm birth rates, fetal birth weight, Aparga score, cesarean rate and so on.

In this study, the investigators will also collect participants' blood samples in first, second and third trimester respectively,and collect cord blood samples, placenta samples,muscle samples and aidpose tissues when they give birh.Thus the investigators can also do some basic reasearch about the potential mechanisms of exercise in preventing GDM.

ELIGIBILITY:
Inclusion Criteria:

* Chinese overweight/obese(prepregnancy BMI≥24kg/m^2) pregnant women aged between 18 years and 45 years with a singleton live fetus.

Exclusion Criteria:

* High-risk pregnancies or diseases that could interfere with participation (or both), such as heart insufficiency, infectious diseases, cervical incompetence, multiple pregnancy,serious blood diseases, serious hypertension,absence of prenatal control, risk of premature labour.
* Prepregnant type 1 or 2 diabetes mellitus.
* Impaired glucose trolerance (IGT) and impaired fasting glucose(IFG)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2014-12; Primary Completion 2016-04 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
the risk of gestational diabetes mellitus | up to 24-28 gestational weeks
  GDM will be diagnosed by an oral glucose tolerance test (OGTT) according to the new World Health Organization criteria as fasting glucose level in fasting whole blood 5.1 mmol/L or more, or 2-hour value 8.5mmol/L or more.Then we can use the rate of GDM ocurrence to represent the risk of gestational diabetes mellitus

SECONDARY OUTCOMES:
weight gain | up to 42 gestatioanl weeks
  use a same scale to measure pregnant women's weight before they give birth,and then subtract their weight prepregnancy. And also, we will use BMI increases as another indicator in representing their weight gain
insulin resistance | up to 13, 26 and 39 gestatioanl weeks
  measure the insulin concentration in the serum of pregnant women in the early(before 13 gestational weeks), mid( between 25-26 gestatianl weeks)and late-term(between 37-39 gestatioanl weeks) of pregnancy, and define their homeostatic model assessments for insulin resistance (HOMA-IR)
adipocytes | up to 13, 26 and 39 gestatioanl weeks
  measure the adipocytes concentrations in the serum of pregnant women in the early(before 13 gestational weeks), mid( between 25-26 gestatianl weeks)and late-term(between 37-39 gestatioanl weeks) of pregnancy, also measure them in the cord blood serum by ELISA.
inflammatory factor | up to 13, 26 and 39 gestatioanl weeks
  measure the inflammatory factor concentrations in the serum of pregnant women in the early(before 13 gestational weeks), mid( between 25-26 gestatianl weeks)and late-term(between 37-39 gestatioanl weeks) of pregnancy, also measure them in the cord blood serum by ELISA.
pregnancy outcome | up to 42 gestational weeks
  collect data about birth weight, Aparga score, duration of pregnancy and delivery mode

CONTACTS AND LOCATIONS:
Overall Officials: Yu-mei Wei, MD, Principal Investigator — Mrs; Chen Wang, PhD, Principal Investigator — Ms
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Halse RE, Wallman KE, Newnham JP, Guelfi KJ. Home-based exercise training improves capillary glucose profile in women with gestational diabetes. Med Sci Sports Exerc. 2014 Sep;46(9):1702-9. doi: 10.1249/MSS.0000000000000302. PMID 24518194
- [Background] Yin YN, Li XL, Tao TJ, Luo BR, Liao SJ. Physical activity during pregnancy and the risk of gestational diabetes mellitus: a systematic review and meta-analysis of randomised controlled trials. Br J Sports Med. 2014 Feb;48(4):290-5. doi: 10.1136/bjsports-2013-092596. Epub 2013 Sep 13. PMID 24037671
- [Background] Tobias DK, Zhang C, van Dam RM, Bowers K, Hu FB. Physical activity before and during pregnancy and risk of gestational diabetes mellitus: a meta-analysis. Diabetes Care. 2011 Jan;34(1):223-9. doi: 10.2337/dc10-1368. Epub 2010 Sep 27. PMID 20876206
- [Background] Kaar JL, Crume T, Brinton JT, Bischoff KJ, McDuffie R, Dabelea D. Maternal obesity, gestational weight gain, and offspring adiposity: the exploring perinatal outcomes among children study. J Pediatr. 2014 Sep;165(3):509-15. doi: 10.1016/j.jpeds.2014.05.050. Epub 2014 Jul 1. PMID 24996985
- [Background] Singh J, Huang CC, Driggers RW, Timofeev J, Amini D, Landy HJ, Miodovnik M, Umans JG. The impact of pre-pregnancy body mass index on the risk of gestational diabetes. J Matern Fetal Neonatal Med. 2012 Jan;25(1):5-10. doi: 10.3109/14767058.2012.626920. Epub 2011 Nov 9. PMID 21955004
- [Background] You T, Arsenis NC, Disanzo BL, Lamonte MJ. Effects of exercise training on chronic inflammation in obesity : current evidence and potential mechanisms. Sports Med. 2013 Apr;43(4):243-56. doi: 10.1007/s40279-013-0023-3. PMID 23494259
- [Background] Golbidi S, Laher I. Exercise induced adipokine changes and the metabolic syndrome. J Diabetes Res. 2014;2014:726861. doi: 10.1155/2014/726861. Epub 2014 Jan 19. PMID 24563869
- [Derived] Wang C, Wei Y, Zhang X, Zhang Y, Xu Q, Su S, Zhang L, Liu C, Feng Y, Shou C, Guelfi KJ, Newnham JP, Yang H. Effect of Regular Exercise Commenced in Early Pregnancy on the Incidence of Gestational Diabetes Mellitus in Overweight and Obese Pregnant Women: A Randomized Controlled Trial. Diabetes Care. 2016 Oct;39(10):e163-4. doi: 10.2337/dc16-1320. No abstract available. PMID 27660125